CLINICAL TRIAL: NCT03994588
Title: Intraperitoneal Polypropylene Light Weight Wide Pore Soft Mesh Versus A. Double Mesh Intraperitoneal Repair for Complex Ventral Hernia: A Prospective Randomized Cohort Study.
Brief Title: Intraperitoneal Polypropylene Light Weight Wide Pore Soft Mesh Repair for Complex Ventral Hernia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Raafat Yahia Afifi, Clinical Professor of General Surgery - primary investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-43-2019
Record Dates: First submitted 2019-06-20; First posted 2019-06-21 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Ventral Hernia
Keywords: Complex ventral hernia; Polypropylene soft mesh; Intraperitoneal repair; Recurrence; Loss of Domain
MeSH Terms: conditions — Hernia, Ventral; Recurrence

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient will be blinded to the study group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study arm (Active Comparator): In this arm a light weight, wide pore, soft polypropylene mesh will be used for intraperitoneal hernia repair
  Interventions: Procedure: Intraperitoneal Mesh hernia repair
- control (Active Comparator): in this arm a double mesh (vicryl + polypropylene mesh) will be used for intraperitoneal hernia repair.
  Interventions: Procedure: Intraperitoneal Mesh hernia repair

INTERVENTIONS:
Procedure: Intraperitoneal Mesh hernia repair — The mesh will be inserted intraperitoneally for complex ventral hernia repair and fixed according the previously described ADMIR technique.

SUMMARY:
Complex ventral hernia is a challenging problem well known to be associated with occurrence of serious complications. The major problems encountered in such cases Include: loss of domain with subsequent increase of intra-abdominal pressure after repair, the huge musculo-fascial defect and skin scarring with possible skin viability problem resulting from the dissection of skin flaps. There is no unified accepted evidence-based approach for its repair and is attended with a high recurrence rate that may reach up to 67%. In a previous study using the ADMIR technique of intraperitoneal repair and after a long-term follow-up the investigator was able to reduce the recurrence rate to 4% after an average follow up period of 142 months. In the current study the investigator will use the same technique of intraperitoneal mesh repair comparing the polypropylene light weight, wide pore, soft mesh with a double mesh using the same polypropylene mesh and a vicryl mesh as a protective layer against the bowel. If it is proven as effective as the mesh with protective layer and with no increased risk of morbidity, this will result in marked reduction of the cost of treatment by nearly 90 % and will abolish the waiting list of patients as the polypropylene mesh is readily available.

DETAILED DESCRIPTION:
According to randomization policy, patients' will be allocated to two groups each one will include 30 subjects: Group I (the study group) in which the investigator will use a polypropylene wide pore soft mesh (Bard, USA). Group II (the control group) in which the investigator will use the same polypropylene mesh in association with Vicryl mesh (Polyglactin 910, VM95, Ethicon, Belgium). The mesh will be prepared by suturing the Vicryl and polypropylene mesh together after folding the edges (2 cm each) and its fixation with four full thickness corners Vicryl 2/0 stay sutures. Another four sutures anchoring the overlapped edges together will be applied at the center of each edge, after that, the mesh will be inserted intraperitoneally in an oblong fashion in defects above the point midway between the umbilicus and symphysis pubis and in horizontal fashion in defects in the hypogastric region with the Vicryl part facing the bowel. U sutures using polypropylene 0 will be applied through the whole thickness of the anterior abdominal wall in order to anchor the four angles of the mesh. Then, the turned over edges of the mesh will be fixed to the inner aspect of the abdominal wall using interrupted full thickness U sutures or mesh stapler (fascia stapler, Medtronic (covidien), USA) according to availability. The same technique will be used in the study group excluding the vicryl mesh. Following mesh fixation, a tailored viable part of the sac will be closed over the mesh to separate it from the subcutaneous tissue in order to minimize seroma formation. Follow-up data will be recorded in a proforma for each patient, noting intraoperative and postoperative complications and postoperative hospital-stay. Each patient will be examined by the surgical team in the Outpatient Clinic at postoperative days 7, 15, and 30 to assess early complications, and at 3 months for one year and every 6 months for 2 years, to assess late complications when necessary after making the scheduled telephone communication.

ELIGIBILITY:
Inclusion Criteria:

Adult patients between 18 and 65 years of age, ASA physical status I - III with complex ventral hernia (defect width above 10 cm, loss of domain above 20 %, recurrent hernia and/or associated with fistula or abdominal wall sinuses).

Exclusion Criteria:

* Age below 18 and above 65 years. The maximum age limit would be 65 years because in our previous studies morbidity was higher in older age group (36, 37).
* Body mass index greater than 45 kg/m2 or weight above 100 kg.
* Pregnancy.
* Associated non treated abdominal malignancy.
* Unstable coronary artery disease, congestive heart failure.
* Significant renal or hepatic impairment;
* Severe bronchopulmonary disease, including chronic obstructive pulmonary disease and obstructive sleep apnea.
* Diabetics with Hb A1c above 7.5.
* Subjects with loss of domain above 20 % who didn't respond to pre-operative progressive pneumoperitoneum.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
The development of persistent abdominal pain (VAS), intestinal obstruction or abdominal wall sinus or fistula formation. | one year
  Manifestations of intestinal obstruction in the form of abdominal pain (VAS), abdominal distention, vomiting and absolute constipation

SECONDARY OUTCOMES:
Hernia recurrence. | three years
  the development of clinically manifest or radiologically detected recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Raafat Y Afifi, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared at the end of the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: one year
Access Criteria: email contact